CLINICAL TRIAL: NCT02880280
Title: Human Menopausal Gonadotropin Combining With Human Chorionic Gonadotropin is Superior to Human Chorionic Gonadotropin in Therapeutic Efficacy in Adolescent Boys With Congenital Hypogonadotropic Hypogonadism
Brief Title: Human Menopausal Gonadotropin Combining With Human Chorionic Gonadotropin Treat Congenital Hypogonadotropic Hypogonadism
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Chunxiu Gong, Professor, Beijing Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BeijingChildrens-01
Record Dates: First submitted 2016-08-11; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Kallmann Syndrome; Hypogonadotropic Hypogonadism
MeSH Terms: conditions — Kallmann Syndrome; Hypogonadism | interventions — Menotropins; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Human Menopausal Gonadotropin (Experimental): Human menopausal gonadotropin contains follicle-stimulating hormone (FSH) and luteinizing hormone (LH)
  Interventions: Drug: Human Menopausal Gonadotropin; Drug: Human Chorionic Gonadotropin
- Human Chorionic Gonadotropin (Experimental): Human chorionic gonadotropin (hCG) is a hormone produced by the embryo after implantation
  Interventions: Drug: Human Chorionic Gonadotropin

INTERVENTIONS:
Drug: Human Menopausal Gonadotropin — Human Menopausal Gonadotropin injection treating congenital hypogonadotropic hypogonadism in teenagers
  Other Names: Human Menopausal Gonadotropin(hMG)
  Arms: Human Menopausal Gonadotropin
Drug: Human Chorionic Gonadotropin — Human Chorionic Gonadotropin injection treating congenital hypogonadotropic hypogonadism in teenagers
  Other Names: Human Chorionic Gonadotropin(hCG)

SUMMARY:
Observe the therapeutic efficacy of human menopausal gonadotropin combining with human chorionic gonadotropin in adolescent boys with congenital hypogonadotropic hypogonadism.

DETAILED DESCRIPTION:
Observe safety and efficacy of human menopausal gonadotropin and human chorionic gonadotropin treating congenital hypogonadotropic hypogonadism in teenagers; which as clinic recommendation, may provide clinical basis for establishing standard treatment guideline in the future. Establish technological process and follow-up precept for human menopausal gonadotropin and human chorionic gonadotropin injection treating congenital hypogonadotropic hypogonadism in teenagers. And find safety and effective dose for teenagers.

ELIGIBILITY:
Inclusion Criteria

Criteria A

* Boy >14yr without any sign of puberty, testis <4ml
* BA ≥12yr
* Sex hormone (LH,FSH, T) are pre-pubertal level
* No other hormones problems (other pituitary glands axis are normal except gonad axis)
* No space occupying lesion, No tumor on MRI of pituitary and hypothalamus area
* Kallmann's syndrome(KS) patients may companies with dysosmia or dysplasia of olfactory bulb or olfactory tract on MRI
* Karyotype is 46，XY
* Exclude chronic diseases, malnutrition

Criteria B

* For the boy <14yr. who companies with micropenis or cryptorchid or hypospadias and they have anosmia or dysplasia of olfactory bulb/olfactory sulcus/olfactory structs on MRI include in.

Criteria C

* As the phenotype of hypogonadotropic hypogonadism are variant, some of them may have partial puberty. So, we enrolled them when they have testis volume >4ml or the testosterone level >200ng/L，companies anosmia or dysplasia of olfactory bulb /olfactory sulcus/ olfactory structs on MRI, and the puberty arrested in half a year. These patients can be diagnosed as Kallmann Syndrome.

Exclusion Criteria:

* Any ascertain reason contributes to the non puberty development (Chromosome abnormal, trauma, surgeries) or any ascertain disease such as Prader-Willi syndrome or hypergonadotropic hypogonadism
* Systemic diseases (such as chronic kidney failure, Mediterranean anemia, poor controlled diabetes)
* Protein-energy malnutrition
* Eating disorder (such as anorexia nervosa, binge eating)
* Any brain diseases history: tumors in brain or pituitary or after their surgeries

Ages: 138 Months to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
testicular volume | Change from Baseline testicular volume at 3 months after treatment

SECONDARY OUTCOMES:
The levels of testosterone serum (It were measured with chemiluminescent immunoassay Elecsys) | Testosterone changes from 3 months onwards after treatment compared to pretreatment

CONTACTS AND LOCATIONS:
Overall Officials: Chunxiu Gong, doctor, Study Director — Beijing Children's Hospital
Locations (1):
- Beijing Children's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Y, Ren XY, Peng YG, Chen SK, Cheng XR, Qin M, Wang XL, Song YN, Fan LJ, Gong CX. Efficacy and safety of human chorionic gonadotropin combined with human menopausal gonadotropin and a gonadotropin-releasing hormone pump for male adolescents with congenital hypogonadotropic hypogonadism. Chin Med J (Engl). 2021 Mar 31;134(10):1152-1159. doi: 10.1097/CM9.0000000000001419. PMID 33813517